CLINICAL TRIAL: NCT00179088
Title: Fiber Metal Taper Prospective Randomized Weight Bearing Investigation
Brief Title: Safety of Non-delayed Weight Bearing After Total Hip Replacement With Non-Cemented Fiber Metal Taper Stem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VUMC IRB#030167; Weight Bearing after THA
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis; Pain
Keywords: Weight-Bearing; Total Hip Replacement; Non-cemented; Randomized; Fiber-Metal-Taper-Stem; Hip; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Pain

INTERVENTIONS:
Behavioral: Patient may be able to put weight on the operated leg

SUMMARY:
The purpose of this study is to determine if full weight bearing following total hip replacement can speed recovery when the hip replacement in the long bone of the leg is not cemented into the bone. When cement is used, most surgeons allow full or nearly full weight bearing following hip replacement. One drawback to cementless implants has been the restriction of weight bearing for six to eight weeks after surgery, during which time patients are allowed to only put their foot flat on the floor of the operated leg without bearing weight on that leg. This study compares the effect of immediate weight bearing on the speed of recovery from hip replacement surgery in two groups of patients receiving a non-cemented total hip replacement: one group is randomly assigned to not bear weight, and the other group is randomly assigned to allowed, tolerated weight bearing from the day of surgery forward.

DETAILED DESCRIPTION:
Patients undergoing non-cemented total hip arthroplasty with a Zimmer Fiber Metal Taper Stem and who meet the inclusion and exclusion criteria are offered the informed consent process. Those consenting are randomized following surgery by flip of a coin into one of two groups: Weight Bearing as Tolerated or Toe Touch Weight Bearing Only. Each patient is followed for two years, and is seen at 6 weeks, 3 months, 1 year and two years. Questionnaires are completed including the Harris Hip Score and the SF-36. Patients complete a compliance survey to determine behavior related to their study group assignment and compliance with their study group. Radiographs are obtained at each post-operative interval and subsidence is evaluated and recorded. Range of motion and ambulation are assessed and recorded also.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* English Speaking
* any form of hip arthritis
* primary total hip arthroplasty
* willing to sign informed consent

Exclusion Criteria:

* under age 18
* non-English speaking
* critically ill patients
* people who are unable to follow-up appropriately due to travel concerns or mental illness.
* revision total hip arthroplasty
* trochanteric osteotomy
* intra-operative fracture
* prisoners
* not willing to sign informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33
Dates: Start 2003-05; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To learn if clinical and radiographic outcomes differ in two groups of patients after THA.

SECONDARY OUTCOMES:
Femoral Stem Subsidence on X-rays at select post-op times.
Return to work status by two years post-operative.
Patient is or is not able to walk without assistive device.
Joint range of motion.
Presence or absence of pain.
Severity of pain if present.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A. Shinar, M.D., Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States